CLINICAL TRIAL: NCT02307266
Title: Effect of Patient Education on Treatment Adherence and Satisfaction Among Acne Patients Receiving Once-daily Epiduo Gel Treatment in Primary Care Clinics
Brief Title: Patient Education in Adherence on Acne (PEAce)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RD.03.SPR.102710
Record Dates: First submitted 2014-11-26; First posted 2014-12-04 (Estimated); Results first posted 2016-09-08 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2016-07

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard of care + supplementary education (Experimental): Subjects will receive supplementary patient educational material in addition to standard-of-care instructions.
  Interventions: Behavioral: Standard of care + supplementary education
- Standard of care (Experimental): Subjects will receive standard-of-care instructions only.
  Interventions: Behavioral: Standard of care
- Standard of care + additional visits (Experimental): Subjects will receive standard-of-care instructions, and two additional clinical visits.
  Interventions: Behavioral: Standard of care + additional visits

INTERVENTIONS:
Behavioral: Standard of care + supplementary education
  Arms: Standard of care + supplementary education
Behavioral: Standard of care + additional visits
  Arms: Standard of care + additional visits
Behavioral: Standard of care
  Arms: Standard of care

SUMMARY:
This is a multi-center, randomised and controlled study in subjects with acne vulgaris. The main objective of this study is to evaluate the effect of a supplementary patient education intervention (in addition to the standard-of-care patient education) on treatment adherence and satisfaction among acne patients receiving once-daily EpiduoTM gel treatment in primary care clinics.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects age of 12 years or older,
2. With facial acne vulgaris that can be managed in primary care

Exclusion Criteria:

1. Female subjects who are pregnant, nursing or planning a pregnancy during the study,
2. Subjects have a very severe variant of acne such as fulminating acne with systemic symptoms (acne fulminans)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United Kingdom (10):
  - Swan Lane Medical Centre, Bolton
  - Burbage Surgery, Burbage
  - South Axholme Practice, Epworth
  - Dr Moss and Partners, Harrogate
  - Barlow Medical Centre, Manchester
  - Leicester Terrace Health Care Centre, Northampton
  - University of Nottingham Health Service, Nottingham
  - Rothwell and Desborough Healthcare Group, Rothwell
  - Albany House Medical Centre, Wellingborough
  - Whitby Group Practice, Whitby

REFERENCES:
- [Derived] Myhill T, Coulson W, Nixon P, Royal S, McCormack T, Kerrouche N. Use of Supplementary Patient Education Material Increases Treatment Adherence and Satisfaction Among Acne Patients Receiving Adapalene 0.1%/Benzoyl Peroxide 2.5% Gel in Primary Care Clinics: A Multicenter, Randomized, Controlled Clinical Study. Dermatol Ther (Heidelb). 2017 Dec;7(4):515-524. doi: 10.1007/s13555-017-0203-4. Epub 2017 Oct 12. PMID 29027127

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care + Supplementary Education: Subjects received supplementary patient educational material in addition to standard-of-care instructions.
- Standard of Care: Subjects received standard-of-care instructions only.
- Standard of Care + Additional Visits: Subjects received standard-of-care instructions, and two additional clinical visits.
Period: Overall Study
Arm/Group | Standard of Care + Supplementary Education | Standard of Care | Standard of Care + Additional Visits
Started | 33 | 33 | 31
Completed | 25 | 32 | 25
Not Completed | 8 | 1 | 6
Not completed — Adverse Event | 3 | 1 | 5
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Lost to Follow-up | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care + Supplementary Education | Standard of Care | Standard of Care + Additional Visits | Total
Number analyzed (Participants) | 33 | 33 | 31 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.1 (9.6) | 21.0 (7.9) | 22.5 (11.1) | 22.5 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 26 | 19 | 67
  Male | 11 | 7 | 12 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 6 | 4 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 29 | 26 | 27 | 82
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Skin Phototype [Number; unit: participants] — Type I: never tan; always sunburn if exposed to sunlight, primarily read headed and lighty complected blondes Type II: frequently burn but are able to tan to a small degree after extended exposure Type III: burn infrequently; tan readily Type IV: rarely burn, tan heavily with moderate sun exposure; esp. Asian, American Indian, Mediterranean and Latin American.
  Type V: have dark constitutive pigmentation, become darker with sun exposure, esp. light complected black individuals, Indian descent.
  Type VI: have the heaviest constitutive pigmentation, esp. dark skinned black individuals.
  participants
    I | 2 | 3 | 2 | 7
    II | 11 | 9 | 11 | 31
    III | 14 | 13 | 12 | 39
    IV | 5 | 6 | 4 | 15
    V | 1 | 2 | 2 | 5
Investigator Global Assessment of Acne [Number; unit: participants] — Clear: Residual hyperpigmentation and erythema may be present Almost clear: a few scattered comedones and a few small papules Mild: Some comedones and some papules and pustules. No nodules present. Moderate: Many comedones, papules and pustules. One nodule may be present. Severe: Covered with comedones, numerous papules and pustules and few nodules may be present.
  Very severe: Highly inflammatory acne covering the face, with nodules present.
  participants
    Almost clear | 8 | 1 | 3 | 12
    Mild | 17 | 22 | 20 | 59
    Moderate | 8 | 10 | 8 | 26
Acne History [Number; unit: participants] — Duration in years
  participants
    Less than 1 year | 12 | 9 | 7 | 28
    Between 1 and 5 years | 11 | 12 | 17 | 40
    More than 5 years | 10 | 12 | 7 | 29

OUTCOME MEASURES:

1. Primary Outcome: Mean Rate of Adherence, as Assessed by Medical Event Monitoring System (MEMS)
Description: To prevent bias, treatment adherence was assessed without subject's knowledge using a Medication Event Monitoring System (MEMS). The treatment was placed in a container fitted with a MEMS cap which recorded the time/date every time it was opened and/or closed. A day with at least one opening was considered a day the subject was adherent. Mean rate of adherence in % corresponds to the number of days the subject was adherent dividided by the total number of days of the study (84 days) times 100.
  Analysis was performed on the "worst-case" population: Missing data were considered as non-adherence.
Time Frame: week 12
Population: Only subjects with usable MEMS data were analyzed, therefore the number of subjects in the analysis population is not the full population.
Measure: Mean (Standard Deviation); unit: percentage of adherence
Arm/Group | Standard of Care + Supplementary Education | Standard of Care | Standard of Care + Additional Visits
Number analyzed (Participants) | 20 | 28 | 23
percentage of adherence | 63.1 (30.2) | 56.5 (24.8) | 48.2 (33.9)
Statistical Analysis 1: Comparison: Standard of Care + Supplementary Education vs Standard of Care; Test type: Superiority or Other; p = 0.3165, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Standard of Care + Supplementary Education vs Standard of Care + Additional Visits; Test type: Superiority or Other; p = 0.0206, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Standard of Care + Supplementary Education | Standard of Care | Standard of Care + Additional Visits
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/31
Other Adverse Events (participants affected / at risk) | 7/33 | 6/33 | 15/31
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care + Supplementary Education (N=33) | Standard of Care (N=33) | Standard of Care + Additional Visits (N=31)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreement covered by contract.